CLINICAL TRIAL: NCT01336920
Title: Phase I Study of Carfilzomib for the Treatment of T-Cell Lymphoma
Brief Title: Carfilzomib in Treating Patients With Relapsed or Refractory T-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0518-10-FB; NCI-2010-02257 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P50CA136411 (NIH); P30CA036727 (NIH)
Record Dates: First submitted 2011-03-23; First posted 2011-04-18 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Peripheral T-cell Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Peripheral; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (carfilzomib) (Experimental): Patients receive carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carfilzomib

INTERVENTIONS:
Drug: carfilzomib — Given IV
  Other Names: Kyprolis; PR-171

SUMMARY:
This phase I trial studies the side effects and best dose of carfilzomib in treating patients with relapsed or refractory T-cell lymphoma. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) of single agent carfilzomib in patients with relapsed and refractory peripheral T-cell lymphoma (PTCL) including angioimmunoblastic T-cell lymphoma (AITL), anaplastic large cell lymphoma (ALCL) anaplastic lymphoma receptor tyrosine kinase (ALK)+/ALK-, adult T-cell leukemia/lymphoma (ATLL), natural killer (NK)-cell lymphoma (NKL), transformed mycosis fungoides (MF) to large cell, and PTCL-unspecified (PTCL-U).

II. To assess the safety and preliminary efficacy of single agent carfilzomib in patients with relapsed and refractory peripheral T-cell lymphoma (PTCL) including angioimmunoblastic T-cell lymphoma (AITL), anaplastic large cell lymphoma (ALCL) ALK+/ALK-, adult T-cell leukemia/lymphoma (ATLL), NK-cell lymphoma (NKL), transformed mycosis fungoides (MF) to large cell, and PTCL-unspecified (PTCL-U).

III. To evaluate nuclear transcription factor kappa-B (NF-kappa B) activation in PTCL tumor tissue and correlate that with response to carfilzomib, a novel proteosome inhibitor, which targets NF-kappa B.

OUTLINE: This is a dose escalation study.

Patients receive carfilzomib intravenously (IV) over 30 minutes on days 1, 2, 8, 9, 15, and 16. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for year 1, then every 4 months for year 2, then every 6 months for years 3 and 4, and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed and refractory PTCL, including angioimmunoblastic T-cell lymphoma (AITL), anaplastic large cell lymphoma (ALCL) ALK+/ALK-, adult T-cell leukemia/lymphoma (ATLL), NK-cell lymphoma (NKL), transformed MF to large cell, and PTCL-unspecified (PTCL-U) patients who have failed standard therapy/transplant for their histological confirmed disease or who are not transplant eligible are eligible to participate in this trial
* Karnofsky performance status >= 70
* ANC >= 700 cells/mm^3, unless due to lymphoma involvement of the bone marrow or spleen
* Platelet count >= 50 mm^3, unless due to lymphoma involvement of the bone marrow or spleen
* Hemoglobin >= 8 g/dL, unless due to lymphoma involvement of the bone marrow
* Liver functions (AST, ALT, bilirubin) =< 3 x upper limits of normal (ULN) unless due to lymphoma or due to Gilberts disease
* Serum creatinine < 2.0 mg/dL or calculated creatinine clearance (CrCl) > 40 mL/min (Cockcroft-Gault)
* LVEF >= 40% 2-D transthoracic ECHO is the preferred method of evaluation; MUGA scan is acceptable if ECHO is not available
* Able to adhere to the study visit schedule and other protocol requirements
* Patients must be willing to give written informed consent, and sign an institutionally approved consent form before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Non-pregnant and non-nursing; men and women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method while on the study
* No serious disease or condition that, in the opinion of the investigator, would compromise the patient's ability to participate in the study
* Patients with a history of coronary artery disease, congestive heart failure, hypertension, diabetes, or hyperlipidemia must have a MUGA or echocardiography, performed within 2 months of study entry

Exclusion Criteria:

* Pregnant or breast feeding females
* Active serious infection requiring treatment within 14 days prior to the start of carfilzomib
* Active hepatitis or uncontrolled HIV
* Unstable angina or myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or EKG evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker
* Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to the start of carfilzomib
* Patients in whom the schedule of oral and IV fluid hydration is contraindicated, e.g., due to pre-existing pulmonary, cardiac, or renal impairment
* Prior malignancies within the past 2 years with exception of adequately treated basal cell, squamous cell skin cancer, or thyroid cancer; carcinoma in situ of the cervix or breast; prostate cancer of Gleason grade 6 or less with stable prostate specific antigen (PSA) levels
* Significant peripheral neuropathy (grades 3-4, or grade 2 with pain) within 14 days prior to the start of carfilzomib
* Known history of allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib)
* Concurrent use of other anti-cancer agents, investigative agents, or treatments
* Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment
* Any other clinically significant medical disease or condition laboratory abnormality or psychiatric illness that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-06-21 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of carfilzomib | 28 days
  MTD of carfilzomib, determined by incidence of dose-limiting toxicity (DLT) as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

OTHER OUTCOMES:
Incidence of adverse events | Up to 30 days after completion of study treatment
  The incidence rates of adverse events will be described by for each dose level. The frequency of occurrence of overall toxicity, categorized by toxicity grades, will be described, assessed by the NCI CTCAE version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Vose, Principal Investigator — University of Nebraska
Locations (3):
- United States (3):
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - University of Nebraska Medical Center, Omaha, Nebraska
  - M D Anderson Cancer Center, Houston, Texas